CLINICAL TRIAL: NCT02856893
Title: APPLE Trial: Feasibility and Activity of AZD9291 (Osimertinib) Treatment on Positive PLasma T790M in EGFR Mutant NSCLC Patients
Brief Title: Osimertinib Treatment on EGFR T790M Plasma Positive NSCLC Patients (APPLE)
Acronym: APPLE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1613; ESR-15-11406 (Other: Astra Zeneca)
Record Dates: First submitted 2016-07-11; First posted 2016-08-05 (Estimated); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: NSCLC
Keywords: AZD9291; Osimertinib; Gefitinib; NSCLC; liquid biopsy; ctDNA
MeSH Terms: interventions — osimertinib; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Osimertinib till progression (Experimental): Osimertinib until PD according to RECIST 1.1
  Interventions: Drug: Osimertinib
- Gefitinib till + blood test/progression than Osimertinib (Experimental): Gefitinib until emergence of positive T790M status ("cfDNA T790M positive progression") followed by Osimertinib until second PD according to RECIST 1.1
  Interventions: Drug: Osimertinib; Drug: Gefitinib
- Gefitinib till progression than Osimertinib (Active Comparator): Gefitinib until PD according to RECIST 1.1 followed by Osimertinib until PD according to RECIST 1.1
  Interventions: Drug: Osimertinib; Drug: Gefitinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib 60 or 40 mg daily until progression
  Other Names: AZD9291, Tagrisso
Drug: Gefitinib — Gefitinib 250mg daily until progression
  Other Names: Iressa
  Arms: Gefitinib till + blood test/progression than Osimertinib; Gefitinib till progression than Osimertinib

SUMMARY:
The phase II APPLE trial gives the opportunity to prospectively validate liquid biopsies as a new standard for testing tumor progression compared with conventional radiological procedure in EGFR mutant advanced NSCLC patients. Moreover based on the sequential T790M test during treatment the investigators will assess the predictive value of liquid biopsies. APPLE trial will examine the best strategy for delivering osimertinib (upfront versus sequential treatment after 1st generation EGFR TKI) in EGFR mutant NSCLC patients. Finally, the trial will also explore the mechanisms of acquired resistance to Osimertinib based on the results of an optional biopsy upon progression.

DETAILED DESCRIPTION:
Primary objective To evaluate the best strategy for delivering Osimertinib (AZD9291) in NSCLC patients with EGFR mutation. The objective is assessed by Progression Free Survival rate at 18 months (PFSR-OSI-18).

Secondary objectives

* To evaluate PFS while receiving osimertinib measured from randomization by RECIST criteria 1.1.
* To evaluate PFS measured from switching to osimertinib by RECIST criteria 1.1.
* To determine the proportion of patients receiving osimertinib based on the determination of cfDNA T790M mutation positive.
* To evaluate PFS-2.
* To evaluate Overall Response Rate (ORR) to osimertinib.
* To evaluate the Treatment duration.
* To evaluate Time to progression (TTP) on osimertinib (measured from switching to osimertinib).
* To evaluate Overall Survival (OS).
* To evaluate brain progression free survival (BPFS).
* Safety.

ELIGIBILITY:
Inclusion:

Registration:

* Pathological diagnosis of adenocarcinoma of the lung carrying common EGFR activating mutations associated with EGFR-TKI sensitivity (Del19 or L858R); performed locally; no other EGFR mutations will be allowed. In case of other (than EGFR) concomitant mutations, discussion with EORTC Headquarters is mandatory;
* Stage IV NSCLC;
* Blood sample available for cfDNA EGFR T790M central testing;
* Age ≥18 years;
* EGFR TKI treatment-naïve eligible to receive first-line treatment with EGFR TKI;
* Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy, investigational agents) if performed more than 12 months before registration;
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations

Randomization:

* Report of adequacy sample for cfDNA EGFR T790M test by central laboratory;
* Prior palliative radiotherapy or surgery are allowed if completed at least 4 weeks before the randomization;
* Patients with brain metastases are allowed provided they are stable (i.e. without evidence of progression by imaging for at least two weeks prior to the first dose of trial treatment and without deterioration of any neurologic symptoms), and have not received steroids for at least 7 days before randomization; Baseline tumor assessment scans are done within 21 days before randomization;
* Evaluable disease as defined below;
* At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have a short axis of ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI), and which is suitable for accurate repeated measurements.
* WHO Performance Status 0-2, with no clinically significant deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks;
* Adequate bone marrow, renal, hepatic and liver function within 21 days from randomization and defined as follows:
* Absolute neutrophil count ≥1.5 x 109/L;
* Platelet count ≥100 x 109/L;
* Haemoglobin ≥9 g/dL;
* Alanine aminotransferase (ALT) ≤2.5x the upper limit of normal (ULN) if no demonstrable liver metastases or ≤5xULN in the presence of liver metastases;
* Aspartate aminotransferase (AST) ≤2.5xULN if no demonstrable liver metastases or ≤5xULN in the presence of liver metastases;
* Total bilirubin ≤1.5xULN if no liver metastases or ≤3xULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases;
* Serum creatinine ≤1.5xULN concurrent with creatinine clearance ≥50 mL/min (measured or calculated by Cockcroft and Gault equation);
* No significant comorbidity that according to the investigator would hamper the participation on the trial;
* Female patients should be using adequate contraceptive measures, should not be breastfeeding, until 12 months after the last dose, and must have a negative pregnancy test (serum or urine) prior to first dose of study drug (within 72 hours); or female patients must have an evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:
* Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
* Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution.
* Documentation of irreversible surgical sterilisation by hysterectomy, bilateraloophorectomy, or bilateral salpingectomy but not tubal ligation.
* Male patients should be willing to use barrier contraception, i.e., condoms

  o Male patients will be advised to arrange for the freezing of sperm samples prior to the start of the study should they wish to father children, and not to donate sperm until 6 months after discontinuation of study treatment." (as per Investigator Brochure, IB)
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Exclusion:

* Treatment with any of the following:
* Prior treatment with any systemic anti-cancer therapy for locally advanced/metastatic NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug;
* Prior treatment with an EGFR-TKI;
* Major surgery (excluding placement of vascular access) within 4 weeks before randomization;
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks before randomization
* Patients currently receiving (or unable to stop use at least 1 week prior to receiving the first dose of study drug) medications or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 (CYP) 3A4;
* Other anti-cancer therapies and alternative medications such as homeopathic treatment, etc;
* Treatment with an investigational drug within five half-lives of the compound or any of its related material, if known;
* Leptomeningeal carcinomatosis; spinal cord compression;
* Any unresolved toxicities from prior systemic therapy (e.g., adjuvant chemotherapy) greater than CTCAE grade 2 at the time of randomization;
* Patients will not be eligible if they have evidence of active malignancy (other than non-melanoma skin cancer or localized cervical cancer or localised and presumed cured prostatic cancer) within 2 years before randomization and are not receiving specific treatment for these malignancies at baseline assessment;
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Active infection will include any patients receiving intravenous treatment for infection; active hepatitis B infection will, at a minimum, include all patients who are Hepatitis B surface antigen positive (HbsAg positive) based on serology assessment. Screening for chronic conditions is not required;
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of Osimertinib or Gefitinib;
* Any of the following cardiac criteria:
* Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 ECGs using local clinic ECG machine-derived QTcF value
* Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec or history of episodes of bradycardia (<50 BPM);
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval.
* Abnormal cardiac function: LVEF < 50% (assessed by MUGA or ECHO)
* Past medical history of ILD (Interstitial Lung Disease), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Dziadziuszko, MD PhD, Principal Investigator — Mecical University of Gdansk, Poland
Locations (23):
- Institut Jules Bordet, Brussels, Bruxelles Région, Belgium
- France (10):
  - Institut Bergonie, Bordeaux
  - CHU de Brest, Brest
  - Centre Francois Baclesse, Caen
  - Centre Hopitalier Intercommunal De Creteil, Créteil
  - Assistance Publique - Hopitaux de Marseille - Hopital Nord, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Centre Paul Strauss, Strasbourg
  - CHU Toulouse - Hopital Larrey, Toulouse
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- King Hussein Cancer Center, Amman, Jordan
- Medical University of Gdansk, Gdansk, Poland
- Slovenia (2):
  - University Clinic Golnik, Golnik
  - The Institute Of Oncology, Ljubljana
- Spain (8):
  - University Hospital A Coruna-Hospital Teresa Herrera, A Coruña
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Institut Catala d'Oncologia - ICO Badalona - Hospital De Mataro, Mataró
  - Virgen del Rocio University Hospital, Seville

REFERENCES:
- [Derived] Remon J, Besse B, Aix SP, Callejo A, Al-Rabi K, Bernabe R, Greillier L, Majem M, Reguart N, Monnet I, Cousin S, Garrido P, Robinet G, Campelo RG, Madroszyk A, Mazieres J, Curcio H, Wasag B, Pretzenbacher Y, Grillet F, Dingemans AC, Dziadziuszko R. Overall Survival From the EORTC LCG-1613 APPLE Trial of Osimertinib Versus Gefitinib Followed by Osimertinib in Advanced EGFR-Mutant Non-Small-Cell Lung Cancer. J Clin Oncol. 2024 Apr 20;42(12):1350-1356. doi: 10.1200/JCO.23.01521. Epub 2024 Feb 7. PMID 38324744

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After registration was completed, eligible patients were randomized within 4 weeks.
Pre-assignment Details: The patients were first registered (step 1) to the trial by authorized sites. The site immediately sent the blood samples for circulating free DNA EGFR T790M (cfDNA T790M) testing to the central lab. Once the sample was assessed (step 2), the site was notified whether they could proceed to patient randomization. Patients were then randomized (step 3) after verification of all eligibility criteria.
Groups:
- Osimertinib Till Progression: Osimertinib until PD according to RECIST 1.1
  Osimertinib: Osimertinib 80 mg daily until progression
- Gefitinib Till + Blood Test/Progression Then Osimertinib: Gefitinib until emergence of positive T790M status ("cfDNA T790M positive progression") or RECIST progression followed by Osimertinib until second PD according to RECIST 1.1
  Gefitinib: Gefitinib 250mg daily until progression Osimertinib: Osimertinib 80 mg daily until second progression
  Note: Osimertinib 60 or 40 mg only upon first progression until second PD
- Gefitinib Till Progression Then Osimertinib: Gefitinib until PD according to RECIST 1.1 followed by Osimertinib until second PD according to RECIST 1.1
  Gefitinib: Gefitinib 250mg daily until progression Osimertinib: Osimertinib 80 mg daily until progression
  Note: Osimertinib 60 or 40 mg only upon first progression until second PD
Period: Overall Study
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Then Osimertinib | Gefitinib Till Progression Then Osimertinib
Started | 53 | 52 | 51
Completed | 20 | 33 | 27
Not Completed | 33 | 19 | 24
Not completed — Lack of Efficacy | 27 | 15 | 19
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Other reasons | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Than Osimertinib | Gefitinib Till Progression Than Osimertinib | Total
Number analyzed (Participants) | 53 | 52 | 51 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 31 | 72
  >=65 years | 32 | 32 | 20 | 84
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [60 to 76] | 69 [61.5 to 75.5] | 61 [54 to 68] | 66 [57 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 39 | 33 | 102
  Male | 23 | 13 | 18 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 40 | 42 | 38 | 120
  More than one race | 6 | 5 | 5 | 16
  Unknown or Not Reported | 5 | 4 | 6 | 15
Region of Enrollment [Number; unit: participants]
  Poland | 1 | 0 | 0 | 1
  Slovenia | 0 | 1 | 1 | 2
  France | 22 | 20 | 21 | 63
  Jordan | 5 | 3 | 7 | 15
  Spain | 25 | 28 | 21 | 74
  Belgium | 0 | 0 | 1 | 1
EGFR mutation [Count of Participants; unit: Participants]
  Del19 | 35 | 33 | 33 | 101
  L858R | 18 | 19 | 18 | 55
Presence of brain metastases [Count of Participants; unit: Participants]
  Yes | 10 | 16 | 14 | 40
  No | 43 | 36 | 37 | 116
WHO Performance Status [Count of Participants; unit: Participants] — Patient's WHO performance status was measured as part of the patient's physical examination. It can take the values ranging from 0 to 4, with 0 denoting a patient "able to carry out all normal activity without restriction" and 4, a patient "Completely disabled; [who] cannot carry on any self-care; totally confined to bed or chair".
  Participants
    0 | 21 | 23 | 26 | 70
    1 | 30 | 28 | 22 | 80
    2 | 2 | 1 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: PFS Rate at 18 Months
Description: The primary endpoint is defined as the proportion of patients at 18 months who are alive and did not experience an event for PFS by RECIST 1.1 while receiving osimertinib (PFS-OSI).
  Specifically, it relates to progression of disease according to RECIST 1.1 or death after switching to osimertinib in arms "Gefitinib till + blood test/progression then Osimertinib" and "Gefitinib till progression then Osimertinib". It is formally assessed in these two arms, whilst only provided as a reference for the "Osimertinib till progression" arm, in which progression of disease or death is measured from baseline considering that patients start with osimertinib.
Time Frame: 18 months after randomization
Population: Per-protocol population defined as patients who have started their study treatment and satisfying all eligibility criteria as per medical review
Measure: Number (84% Confidence Interval); unit: Percentage of participants
Groups:
- Osimertinib Till Progression: Osimertinib until PD according to RECIST 1.1
  Osimertinib: Osimertinib 80 mg daily (QD) until progression
- Gefitinib Till + Blood Test/Progression Than Osimertinib: Gefitinib until emergence of positive T790M status ("cfDNA T790M positive progression") followed by Osimertinib until second PD according to RECIST 1.1
  Osimertinib: Osimertinib 80 mg daily (QD) mg daily until progression
  Gefitinib: Gefitinib 250mg daily until progression
- Gefitinib Till Progression Than Osimertinib: Gefitinib until PD according to RECIST 1.1 followed by Osimertinib until PD according to RECIST 1.1
  Osimertinib: Osimertinib 80 mg daily (QD) until progression
  Gefitinib: Gefitinib 250mg daily until progression
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Than Osimertinib | Gefitinib Till Progression Than Osimertinib
Number analyzed (Participants) | 45 | 47 | 44
Percentage of participants | 51.1 [40.2 to 61.0] | 67.2 [56.4 to 75.9] | 53.5 [42.3 to 63.5]
Statistical Analysis 1: Comparison: Gefitinib Till + Blood Test/Progression Than Osimertinib; Each arm will be assessed individually against a historical control with a single proportion test. The test is designed to reject a PFS rate at 18 months of 40% (null hypothesis) at the 0.08 significance level. Under the alternative hypothesis of a PFS rate at 18 months of 60%, 49 patients are required to reach a power of 84%; Test type: Other — The decision rule is based on confidence intervals. The treatment strategy will be considered feasible (H0 is rejected) if the lower bound of the 84% two-sided confidence interval of the PFS rate at 18 months is greater than 40%; Kaplan-Meier survival rate = 67.2, 84% CI 2-sided [56.4 to 75.9] — The population parameter is PFS Rate at 18 months in the "Gefitinib till + blood test/progression then Osimertinib" arm. The decision rule is based on the lower bound of the estimated confidence interval around the point estimate
Statistical Analysis 2: Comparison: Gefitinib Till Progression Than Osimertinib; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Kaplan-Meier survival rate = 53.5, 84% CI 2-sided [42.3 to 63.5] — The population parameter is PFS Rate at 18 months in the "Gefitinib till progression than Osimertinib" arm. The decision rule is based on the lower bound of the estimated confidence interval around the point estimate

2. Secondary Outcome: PFS While Receiving Osimertinib by RECIST Criteria 1.1
Description: For patients in arm "Osimertinib till progression", progression Free Survival "while receiving osimertinib" (PFS-OSI) is defined as the time interval between the date of randomization and the date of disease progression according to the RECIST 1.1 or death whichever comes first.
  For patients in arm "Gefitinib till + blood test/progression than Osimertinib" and "Gefitinib till progression than Osimertinib "switching to osimertinib, PFS-OSI is defined as the time interval between the date of randomization and the date of disease progression or death "after switching to osimertinib" whichever comes first. For patients in those two arms who do not start osimertinib for any reason, PFS-OSI is defined as the time interval between the date of randomization and the date of first disease progression according to the RECIST 1.1 or death whichever comes first.
  The median will be calculated using the Kaplan-Meier method.
Time Frame: From randomization till the date of progression on osimertinib or death, an average of 2 years.
Population: Per-protocol population defined as patients who started treatment and satisfied all eligibility criteria as per medical review.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gefitinib Till + Blood Test/Progression Than Osimertinib: Gefitinib until emergence of positive T790M status ("cfDNA T790M positive progression") followed by Osimertinib until second PD according to RECIST 1.1
  Osimertinib: Osimertinib 80 mg daily (QD) until progression
  Gefitinib: Gefitinib 250mg daily until progression
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Than Osimertinib | Gefitinib Till Progression Than Osimertinib
Number analyzed (Participants) | 45 | 47 | 44
months | 19.48 [14.42 to 26.97] | 21.98 [18.56 to NA] — upper limit for the confidence interval around the median was not reached due to an insufficient number of participants with event | 20.17 [14.62 to 34.99]

3. Secondary Outcome: Proportion of Patients Receiving Osimertinib Based on the Determination of cfDNA T790M Mutation Positive
Description: The proportion of patients receiving osimertinib based on the determination of cfDNA T790M is the number of patients receiving at least 1 dose of osimertinib based on the determination of cfDNA T790M (positive mutation). This endpoint is only defined and applicable for the "Gefitinib till + blood test/progression than Osimertinib" arm.
  The 95% confidence intervals will be calculated using the exact binomial method.
Time Frame: From randomization till the date of positive cfDNA T790M status or death, on average 2 years.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Gefitinib Till + Blood Test/Progression Than Osimertinib
Number analyzed (Participants) | 47
proportion of participants | 0.170 [0.076 to 0.308]

4. Secondary Outcome: Time to Progression on Osimertinib
Description: Time to progression on osimertinib is defined as the time interval between the date receiving osimertinib and the date of disease progression. Death is not counted as an event. If the event has not been observed or if the patient dies before the analysis cut-off date, then the patient is censored at the date of the last disease assessment or the date of death prior the cut-off date. Patients not receiving osimertinib are excluded for this endpoint. The nature of this endpoint is different in Arm "Osimertinib till progression" (first line progression) compared to the other two arms (second line progression).
Time Frame: From randomization till the date of progression on osimertinib or death, on average 2 years.
Population: Per-protocol population defined as patients who started treatment and satisfied all eligibility criteria as per medical review. Only patients who started osimertinib are included in this analysis.
Measure: Median (95% Confidence Interval); unit: Time in months
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Than Osimertinib | Gefitinib Till Progression Than Osimertinib
Number analyzed (Participants) | 45 | 31 | 34
Time in months | 19.48 [14.42 to 32.53] | 10.81 [8.15 to 15.57] | 7.39 [5.32 to 11.63]

5. Secondary Outcome: Overall Response Rate (ORR) to Osimertinib
Description: Overall response rate (ORR) to osimertinib is defined as the proportion of patients achieving complete response (CR) or partial response (PR) during osimertinib treatment.
  The analysis of overall response rate (ORR) on osimertinib was performed on the per-protocol population. Patients not receiving Osimertinib will not be included in the osimertinib analysis.
Time Frame: Time from randomization until end of osimeritinib treatment, or death, on average 2 years.
Population: Per-protocol population defined as patients who started treatment and satisfied all eligibility criteria as per medical review. Patients not receiving Osimertinib will not be included in the osimertinib analysis.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Than Osimertinib | Gefitinib Till Progression Than Osimertinib
Number analyzed (Participants) | 45 | 32 | 34
proportion of patients | 0.889 [0.759 to 0.963] | 0.656 [0.468 to 0.814] | 0.588 [0.407 to 0.754]

6. Secondary Outcome: Treatment Duration
Description: treatment duration is measured from randomization till the last day of treatment administration. For patients in arm "Osimertinib till progression" this corresponds to the whole osimertinib treatment duration, and for patients in the other two arms, to the whole gefitinib and osimertinib treatment duration. Patients for whom no end of treatment form has been collected, are known be alive and have not started any off protocol treatment prior to clinical cut off date will be considered as still on treatment and censored in this analysis.
Time Frame: From randomization till the date of end of protocol treatment
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Than Osimertinib | Gefitinib Till Progression Than Osimertinib
Number analyzed (Participants) | 45 | 47 | 44
Months | 24.4 [16.6 to 28.0] | 21.6 [14.7 to 25.6] | 16.2 [12.0 to 27.2]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time interval between the date of randomization and the date of death from any cause. Patients still alive at the analysis cut-off date are censored at the last date known to be alive (before the cut-off date).
  The median will be calculated using the Kaplan-Meier method.
Time Frame: From randomization till the date of death
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Than Osimertinib | Gefitinib Till Progression Than Osimertinib
Number analyzed (Participants) | 45 | 47 | 44
Months | NA [28.40 to NA] — Median and upper limit could not be determined due to an insufficient number of participants with events | NA [26.40 to NA] — Median and upper limit could not be determined due to an insufficient number of participants with events | 42.84 [27.01 to NA] — upper limit could not be determined due to an insufficient number of participants with events

8. Secondary Outcome: Brain Progression Free Survival (BPFS)
Description: Brain progression free survival is defined as the time interval between the randomization and the date of brain progression (progression within target lesions in the brain, unequivocal progression in non-target lesions in the brain, or appearance of new lesions in the brain) or death whichever comes first.
  CT scan will be used to evaluate new or recurrence progression in the brain. If the event has not been observed or if the patient dies or has PD that hampered further assessment/evaluation of brain progression, then the patient is censored at the date of the last follow up examination.
  The medians have been estimated using the Kaplan-Meier method.
Time Frame: From randomization till the date of progression in the brain
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Than Osimertinib | Gefitinib Till Progression Than Osimertinib
Number analyzed (Participants) | 45 | 47 | 44
Months | 34.30 [25.00 to NA] — Upper limit could not be determined due to an insufficient number of participants with events | 24.44 [17.87 to 28.58] | 21.39 [14.49 to 42.84]

9. Secondary Outcome: PFS-2
Description: In the "Osimertinib till progression" arm, PFS-2 is calculated as the time between randomization and the second PD by RECIST 1.1 or death, irrespective of treatment(s) received.
  In the other two arms, PFS-2 is calculated as the time between randomization and the second PD by RECIST 1.1 or death after switching to osimertinib, the first PD being PD by RECIST 1.1 or by positive cfDNA T790M status. For patients unable to start osimertinib, PFS-2 is calculated as the time between randomization and the second PD by RECIST 1.1 on any subsequent off protocol anticancer treatment line.
  If no PFS-2 event has been observed prior to the analysis cut-off date, then the patient is censored at the date of the last disease assessment before the cut-off date.
Time Frame: From randomization till the date of second progression on second line treatment
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Than Osimertinib | Gefitinib Till Progression Than Osimertinib
Number analyzed (Participants) | 45 | 47 | 44
Months | 25.76 [21.78 to NA] — Upper limit could not be determined due to an insufficient number of participants with events | 21.98 [18.56 to NA] — Upper limit could not be determined due to an insufficient number of participants with events | 20.27 [14.82 to 34.99]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during a 3 year and 9 months period.
Arm/Group | Osimertinib Till Progression | Gefitinib Till + Blood Test/Progression Than Osimertinib | Gefitinib Till Progression Than Osimertinib
All-Cause Mortality (participants affected / at risk) | 19/53 | 20/52 | 18/51
Serious Adverse Events (participants affected / at risk) | 9/53 | 6/52 | 13/51
Other Adverse Events (participants affected / at risk) | 52/53 | 51/52 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osimertinib Till Progression (N=53) | Gefitinib Till + Blood Test/Progression Than Osimertinib (N=52) | Gefitinib Till Progression Than Osimertinib (N=51)
ACUTE RESPIRATORY INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
BILATERAL RENAL INFARCTS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
DECREASE ORAL INTAKE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
DETERIORATION OF HEALTH STATUS (General disorders) | 0 (0) | 0 (0) | 1 (3)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INFECTED SKIN ULCER IN THE RIGHT LEG (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
LUNG INFECTION (PNEUMONIA) (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
ORAL MUCOSITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SPLENIC INFARCT (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INTRAEPITHELIAL CECAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PULMONARY INFECTION (PNEUMOCOCCAL PNEUMONIA) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ACUTE GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LEPTOMENINGEAL CARCINOMATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MULTIORGAN FAIL (General disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL INSUFFICIENCY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
SEGMENTAL KINETIC DISORDERS OF THE LEFT VENTRICULE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
SEPTIC SHOCK (URINARY INFECTION) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SEVERE SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
RIGHT PLEURAL SPILL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
NEUROLOGICAL TROUBLES (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
DECREASE LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osimertinib Till Progression (N=53) | Gefitinib Till + Blood Test/Progression Than Osimertinib (N=52) | Gefitinib Till Progression Than Osimertinib (N=51)
Anemia (Blood and lymphatic system disorders) | 10 (10) | 10 (10) | 5 (5)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2) | 3 (3) | 3 (3)
Dry Eye (Eye disorders) | 1 (1) | 6 (6) | 7 (7)
Other adverse events (Eye disorders) | 1 (1) | 4 (4) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 6 (6) | 6 (6)
Constipation (Gastrointestinal disorders) | 7 (7) | 6 (6) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 27 (27) | 30 (30) | 28 (28)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 5 (5) | 6 (6)
Hemorrhoids (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 7 (7) | 9 (9) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 8 (8) | 8 (8)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (4)
Other adverse events (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 4 (4) | 0 (0)
Edema Limbs (General disorders) | 2 (2) | 2 (2) | 4 (4)
Fatigue (General disorders) | 18 (18) | 17 (17) | 15 (15)
Fever (General disorders) | 3 (3) | 2 (2) | 3 (3)
Flu Like Symptoms (General disorders) | 1 (1) | 1 (1) | 3 (3)
Non-Cardiac Chest Pain (General disorders) | 6 (6) | 2 (2) | 7 (7)
Pain (General disorders) | 5 (5) | 4 (4) | 7 (7)
Other adverse events (Hepatobiliary disorders) | 0 (0) | 0 (0) | 5 (5)
Lung Infection (Infections and infestations) | 1 (1) | 3 (3) | 3 (3)
Nail Infection (Infections and infestations) | 4 (4) | 4 (4) | 3 (3)
Papulopustular Rash (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Paronychia (Infections and infestations) | 7 (7) | 7 (7) | 8 (8)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Rhinitis Infective (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 2 (2) | 5 (5) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 6 (6) | 5 (5)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 7 (7) | 5 (5)
Other adverse events (Infections and infestations) | 8 (8) | 5 (5) | 4 (4)
Other adverse events (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 7 (7) | 14 (14) | 15 (15)
Alkaline Phosphatase Increased (Investigations) | 4 (4) | 3 (3) | 5 (5)
Aspartate Aminotransferase Increased (Investigations) | 5 (5) | 12 (12) | 13 (13)
Blood Bilirubin Increased (Investigations) | 0 (0) | 2 (2) | 4 (4)
Cholesterol High (Investigations) | 2 (2) | 3 (3) | 2 (2)
Cpk Increased (Investigations) | 2 (2) | 1 (1) | 3 (3)
Creatinine Increased (Investigations) | 3 (3) | 5 (5) | 3 (3)
Electrocardiogram Qt Corrected Interval (Investigations) | 4 (4) | 3 (3) | 2 (2)
Ggt Increased (Investigations) | 6 (6) | 3 (3) | 4 (4)
Neutrophil Count Decreased (Investigations) | 6 (6) | 3 (3) | 4 (4)
Platelet Count Decreased (Investigations) | 12 (12) | 7 (7) | 2 (2)
Weight Gain (Investigations) | 5 (5) | 4 (4) | 10 (10)
Weight Loss (Investigations) | 19 (19) | 15 (15) | 19 (19)
White Blood Cell Decreased (Investigations) | 3 (3) | 3 (3) | 0 (0)
Other adverse events (Investigations) | 2 (2) | 3 (3) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 12 (12) | 11 (11) | 9 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 8 (8) | 10 (10)
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 6 (6)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 6 (6)
Neck Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 5 (5)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 5 (5)
Dizziness (Nervous system disorders) | 2 (2) | 8 (8) | 4 (4)
Dysgeusia (Nervous system disorders) | 7 (7) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 10 (10) | 11 (11)
Paresthesia (Nervous system disorders) | 4 (4) | 3 (3) | 3 (3)
Other adverse events (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 6 (6)
Depression (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 3 (3)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0)
Cystitis Noninfective (Renal and urinary disorders) | 1 (1) | 1 (1) | 5 (5)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (9) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 3 (3) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4)
Other adverse events (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 22 (22) | 18 (18) | 17 (17)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 3 (3)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Nail Loss (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 10 (10) | 10 (10)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 11 (11) | 24 (24) | 19 (19)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7) | 5 (5)
Other adverse events (Skin and subcutaneous tissue disorders) | 9 (9) | 11 (11) | 6 (6)
Hypertension (Vascular disorders) | 7 (7) | 8 (8) | 5 (5)
Thromboembolic Event (Vascular disorders) | 7 (7) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results. There are no timeline for this review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT02856893/Prot_SAP_000.pdf